CLINICAL TRIAL: NCT06633055
Title: A Phase I Clinical Trial of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JH013 Injection in Healthy Subjects
Brief Title: A Phase I Clinical Trial of JH013 Injection
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BPL-JH013-HV-1001
Record Dates: First submitted 2024-09-28; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Healthy Subjects (HS)
Keywords: Dose escaltion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- JH013 injections 75mg (Experimental): 6 subjects receive JH013 at a dose of 75 mg and 2 subjects receive the same volume placebo
  Interventions: Drug: JH013 injection; Drug: Placebo
- JH013 injections 150mg (Experimental): 6 subjects will receive JH013 injections 150mg，2 subjects receive the same volume placebo
  Interventions: Drug: JH013 injection; Drug: Placebo
- JH013 injections 300mg (Experimental): 6 subjects receive JH013 at a dose of 300 mg and 2 subjects receive the same volume placebo
  Interventions: Drug: JH013 injection; Drug: Placebo
- JH013 injections 500mg (Experimental): 6 subjects receive JH013 at a dose of 500 mg and 2 subjects receive the same volume placebo
  Interventions: Drug: JH013 injection; Drug: Placebo

INTERVENTIONS:
Drug: JH013 injection — JH013 injection is a BAFF-R inhibitor monoclonal antibody
  Other Names: JH013
Drug: Placebo — JH013 injections placebo
  Other Names: JH013 Placebo

SUMMARY:
This is a phase I clinical trial with a single dose escalation to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of JH013 injection in healthy subjects

DETAILED DESCRIPTION:
Four dose groups were set up, 75 mg, 150 mg, 300 mg, and 500 mg, respectively. Eight subjects (6 subjects received JH013 injection, 2 subjects received placebo) were planned to be included in each dose group for subcutaneous administration.The safety and tolerability within 48 hours after administration were first observed in each dose group with 2 subjects (1 subject receiving JH013 injection and 1 subject receiving placebo),after that, the remaining 6 subjects (5 receiving JH013 injection and 1 receiving placebo) were enrolled. Each subject may only participate in this trial in one dose group, and the next higher dose trial will only be allowed after it has been determined that the previous dose has been well safe and tolerated within 28 days of dosing (as determined by an independent, unblinded third-party physician in conjunction with the investigator and sponsor). When the safety evaluation meets the termination criteria during the dose escalation process, the dose between the dose group and the previous dose group can be returned if necessary after discussion by the investigator and the sponsor, and the maximum safe tolerated dose can be explored again. When the dose is escalated to the highest dose set by the protocol and the dose termination criteria are not met, it is up to the investigator and the sponsor to discuss whether to expand to a higher dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female aged 18-55 years (age including cut-off values);
* There were no abnormalities in clinically significant vital signs, physical examination, laboratory tests, and 12-lead ECG;
* Weight ≥ 50 kg for males and ≥45 kg for females; Body mass index (BMI) between 18.0 and 26 kg/m2 (including cut-off values, body mass index = weight/height2);
* Females of potential childbearing potential with a negative blood β-HCG test within 72 hours prior to dosing (postmenopausal women who have amenorrhea for at least 12 months are considered non-childbearing and women who are known to have undergone hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or ligation, and a pregnancy test is not required);
* Subjects understand and comply with the study process, participate voluntarily, and sign the informed consent form

Exclusion Criteria:

* Subject has a history of malignancy prior to screening, or has been screened for malignancy, and the possibility of malignancy cannot be reasonably ruled out
* Subject has a history of autoimmune disease prior to screening
* γ interferon release assay results ≥ 2 times the upper limit of normal
* Any history of infection requiring hospitalization or receiving antivirals, antibiotics, antifungals, antiparasitic drugs, or vaccinations within 4 weeks prior to the application of the study drug
* Those who have positive test results for human immunodeficiency virus (HIV) antibody, hepatitis B virus (HBV) surface antigen, hepatitis C virus (HCV) antibody or syphilis antibody
* Patients with a history of previous and/or current heart disease (including New York Heart Association Class III/IV heart failure), gastrointestinal, renal, endocrine, neurological, autoimmune, hematologic (including pancytopenia, aplastic anemia or anaemia, etc.), metabolic (including diabetes), severe lung disease and psychiatric illness
* History of organ transplantation: such as heart, lung, kidney, liver, or hematopoietic stem cell transplantation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety metrics | from Administration to Day57.
  Including Adverse events defined by CTCAE 5.0（Common Terminology Criteria for Adverse Events Version 5.0) Version 5.0）

SECONDARY OUTCOMES:
t1/2 | from Administration to Day57.
  Half-life
Cmax | from Administration to Day57.
  maximum plasma concentration
CD45+CD19+ B cell | from Administration to Day57.
  Detection CD45+CD19+ B cell count and ratio in blood
B cell activation factor (BAFF) | from Administration to Day57.
  Detection B cell activation factor (BAFF) in serum
JH013 antibody | from Administration to Day57.
  Detection of JH013 antibody occupancy in serum
CD45+CD3+T cell | from Administration to Day57.
  Detection of CD45+CD3+T cell count and ratio blood
Drug immunogenicity | from Administration to Day57.
  Detection of anti-drug antibodies in serum

CONTACTS AND LOCATIONS:
Overall Officials: chen Rui, Dr, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No